CLINICAL TRIAL: NCT03152929
Title: Paravertebral Block Versus Pectoral Nerve Block for Analgesia Following Mastectomy
Brief Title: Paravertebral Block (PVC) Versus Pectoral Nerve Block (PEC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Standards of care changed at the institution so that PEC procedures were no longer common or preferred as a method of pain control for breast surgery.
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-306
Record Dates: First submitted 2017-03-01; First posted 2017-05-15 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Surgery; Breast; Pectoral Nerve Block; Paravertebral Block; Analgesia; Mastectomy
MeSH Terms: conditions — Breast Neoplasms; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two interventional arms (paravertebral block versus pectoral nerve block).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paravertebral Block (Active Comparator): The Paravertebral Block is performed along the spine utilizing ultrasound guided technique (20-30 mL 0.5% Ropivacaine)
  Interventions: Drug: Paravertebral Block
- Pectoral Nerve Block (Active Comparator): The Pectoral Nerve Block is performed anteriorly, at the level of the axillary line, also utilizing ultrasound guided technique (20-30 mL 0.5% Ropivacaine)
  Interventions: Drug: Pectoral Nerve Block

INTERVENTIONS:
Drug: Paravertebral Block — 20-30 mL 0.5% Ropivacaine
  Other Names: PVB
  Arms: Paravertebral Block
Drug: Pectoral Nerve Block — 20-30 mL 0.5% Ropivacaine
  Other Names: PEC
  Arms: Pectoral Nerve Block

SUMMARY:
The purpose of this study is to compare two standard methods of pain control management used at Spectrum Health for patients undergoing breast surgery. The two methods being compared are the paravertebral block (PVB) and the pectoral nerve block (PEC). Postoperative pain control is essential following any major operative procedure. A variety of methods have been used to ensure adequate pain control, each with its own advantages and risks. Increasingly, attention has focused on regional methods of analgesia, which may allow for reduction in systemic narcotic use and their associated complications. Proposed benefits of regional analgesia and a resultant reduction in narcotic use include decreased risk of cancer progression, decreased length of stay, and decreased risk of ileus.

DETAILED DESCRIPTION:
The purpose of this study is to compare the clinical profiles of two currently acceptable analgesia techniques. The most common regional block used to achieve postoperative analgesia following mastectomy is the paravertebral block, during which local anesthetic is injected into the paravertebral space which contains the thoracic spinal nerves, between the costotransverse ligament and the pleura. At our institution there has been recent interest in an alternative regional block. The pectoral nerve block is performed by injecting anesthetic between the pectoralis major and the pectoralis minor (PECs I) or between the pectoralis minor and the serratus anterior (PEC II).

The proposed advantage of the pectoral nerve block for regional anesthesia during breast surgery is equal analgesic efficacy with fewer potential complications.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years of age
* Total mastectomy or partial mastectomy with or without reconstruction OR planned lumpectomy.
* Patient determined by their surgeon as medically able to receive a regional block for post-operative analgesia
* Patient agrees to participate in the study and signs informed consent

Exclusion Criteria:

* Neoadjuvant radiation therapy
* Stage IV cancer
* Previous breast surgery (excluding percutaneous biopsies of all types)
* History of either PVB or PEC procedures
* Planned general anesthesia use during surgery
* Allergies to ropivacaine, midazolam, fentanyl, or propofol
* Pregnant women
* Prisoners
* Adults unable to consent
* Non-English-speaking patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Melink, MD, Principal Investigator — Corewell Health West
Locations (1):
- Esther L Peariso, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: enrollment was stopped prematurely as the Standard of Care changed due to rising evidence during the enrollment period.
Period: Overall Study
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Started | 40 | 49
Completed | 40 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paravertebral Block | Pectoral Nerve Block | Total
Number analyzed (Participants) | 40 | 49 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.15 (10.18) | 64.24 (11.42) | 64.65 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 49 | 89
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 39 | 48 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 49 | 89

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Narcotic Use
Description: Participants for whom Narcotics were used for pain during surgery
Time Frame: intraoperatively, average of about 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 40 | 49
Participants | 26 | 29

2. Primary Outcome: Post Anesthesia Care Unit (PACU) Narcotic Use
Description: Participants for whom Narcotics were used in PACU
Time Frame: in PACU, generally 1-3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 40 | 49
Participants | 20 | 33

3. Primary Outcome: Postoperative Narcotic Use
Description: Participants for whom Narcotics were used postoperatively
Time Frame: First 24 hours post-PACU (or until discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 40 | 49
Participants | 3 | 1

4. Secondary Outcome: Pain Control Measured by Length of Operation
Description: Measuring pain control by how long (in minutes) patient is in surgery
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 40 | 49
minutes | 61.80 (16.42) | 64.14 (20.20)

5. Secondary Outcome: Pain Control Measured by Estimated Blood Loss
Description: Measuring blood loss (in ml) during surgery
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 40 | 49
milliliters | 10.85 (8.3) | 13.8 (12.29)

6. Secondary Outcome: Participants With Postoperative Nausea
Description: count of participants who reported nausea after surgery
Time Frame: 2 weeks postoperative
Population: Paravertebral population had one non-reporting participant
Measure: Count of Participants; unit: Participants
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 39 | 49
Participants | 0 | 1

7. Secondary Outcome: Pain Control Measured by Pain Scale
Description: Pain measured on scale of one to ten, one being least amount of pain and ten the greatest.
Time Frame: 2 weeks postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 40 | 49
score on a scale | 2 (1.33) | 2.4 (1.4)

8. Secondary Outcome: Pain Control Measured by the Use of Pain Pills Postoperatively
Description: Participants who used narcotic pain pills postoperatively
Time Frame: 2 weeks postoperative
Population: Paravertebral Block arm had one participant with no response
Measure: Count of Participants; unit: Participants
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 39 | 49
Participants | 20 | 24

9. Secondary Outcome: Pain Control Measured by Calls to Physicians Office Relating to Pain
Description: Number of phone calls made to physician office regarding pain
Time Frame: 2 weeks postoperative
Population: one participant in each arm did not have a response recorded
Measure: Count of Participants; unit: Participants
Arm/Group | Paravertebral Block | Pectoral Nerve Block
Number analyzed (Participants) | 39 | 48
Participants
  no phone calls to physician office regarding pain | 38 | 44
  1 phone call to physician office regarding pain | 1 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of surgery until the 2 week post op appointment
Description: pain was not considered an adverse event unless it reached a grade 3 by CTCAE v4.0
Arm/Group | Paravertebral Block | Pectoral Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/49
Other Adverse Events (participants affected / at risk) | 0/40 | 0/49

LIMITATIONS AND CAVEATS:
Study was terminated early due to clinical practice outpacing the science of the trial. At the time of stopping enrollment, pectoral nerve blocks were being used standardly. Therefore, we could not ethically continue to randomize patients to both arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT03152929/Prot_SAP_000.pdf